CLINICAL TRIAL: NCT01371331
Title: A Multicentre, Open-label, Pharmacokinetic Study of Modigraf® (Tacrolimus Granules) in de Novo Paediatric Allograft Recipients
Brief Title: A Study to Determine Pharmacokinetics of Children Receiving Modigraf (Tacrolimus Granules) Following Solid Organ Transplantation
Acronym: OPTION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Europe Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: F506-CL-0403; 2009-012258-19 (EudraCT Number)
Record Dates: First submitted 2011-06-09; First posted 2011-06-10 (Estimated); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Kidney Transplantation; Heart Transplantation; Liver Transplantation
Keywords: Kidney Transplantation; Pharmacokinetics; Heart Transplantation; Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tacrolimus granules (Experimental): oral
  Interventions: Drug: Tacrolimus granules

INTERVENTIONS:
Drug: Tacrolimus granules — oral
  Other Names: Modigraf

SUMMARY:
The purpose of this study is to find out how much of Modigraf is absorbed and used in the body and how fast it leaves the body (Pharmacokinetics). The results will then help to decide how much Modigraf in future can be given safely to children and young people following transplantation.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the pharmacokinetics (PK) of tacrolimus following oral administration of Modigraf, after the first oral dose and at steady state in paediatric subjects undergoing de novo allograft transplantation.

ELIGIBILITY:
Inclusion Criteria:

* The subject is the recipient of a solid organ (liver, kidney or heart) transplant. Multiorgan transplants are acceptable as long as one of the organs transplanted is liver, kidney or heart

Exclusion Criteria:

* The subject has previously received another organ transplant (including liver, kidney or heart re-transplantation)
* Subject has a high immunological risk, defined as a Panel Reactive Antibody (PRA) score >50% in the previous 6 months (only applicable for renal transplant recipients)
* Cold ischemia time of the donor kidney greater than 30 hours (only applicable for renal transplant recipients)
* Subject receives an AB0 incompatible donor organ
* Subject has significant renal impairment, defined as having serum creatinine ≥230 μmol/l (≥2.6 mg/dl) pre-transplantation (not applicable for renal transplant recipients)
* Subject has significant liver disease, defined as having elevated Alanine Aminotransferase (ALT) and/or Asparate Aminotransferase (AST) and/or Total Bilirubin levels 3 times the upper value of the normal range during the 28 days prior to transplantation (not applicable for liver transplant recipients)
* Subject with pulmonary vascular resistance greater than 4 Wood units which is unresponsive to treatment
* Subjects with malignancies or a history of malignancy within the last 5 years
* Subject has a significant, uncontrolled systemic infection and/or severe diarrhea, vomiting, active upper gastrointestinal disorder that may affect the absorption of tacrolimus or has an active peptic ulcer
* Subject requires systemic immunosuppressive medication for any indication other than transplantation
* Recipient or donor known to be HIV, HCV or HBV positive
* Known allergy or intolerance to steroids, macrolide antibiotics, basiliximab or tacrolimus
* Subject is currently participating in another clinical trial and/or has been taking an investigational drug in the 3 months prior to transplantation
* Subject is unlikely to comply with the visits scheduled in the protocol
* Subjects taking or requiring to be treated with medication or substances prohibited by this protocol

Ages: 0 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2011-06-09 (Actual); Primary Completion 2015-02-03 (Actual); Study Completion 2015-02-03 (Actual)

PRIMARY OUTCOMES:
Determine AUCtau (area under the plasma concentration-time curve for a dosing interval) | on Day 1 and Day 7 (+/- 7 days)
Determine Cmax (maximum concentration) | on Day 1 and Day 7 (+/- 7 days)
Determine tmax (time to attain Cmax) | on Day 1 and Day 7 (+/- 7 days)
Determine Ctrough (plasma concentration at the end of a dosing interval) | on Day 1 and Day 7 (+/- 7 days)

SECONDARY OUTCOMES:
Rejection episodes | 14 days
Patient survival | 14 days
Graft survival | 14 days
Assessment of safety through the evaluation of Adverse Events, laboratory parameters and vital signs | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Senior Study Manager, Study Chair — Astellas Pharma Europe Ltd.
Locations (10):
- Site 40, Brussels, Belgium
- Site: 60, Bron, France
- Germany (2):
  - Site 31, Hanover
  - Site 30, Heidelberg
- Site 50, Warsaw, Poland
- Spain (3):
  - Site 22, Madrid
  - Site 20, Madrid
  - Site 21, Madrid
- United Kingdom (2):
  - Site 10, Birmingham
  - Site 13, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Webb NJA, Baumann U, Camino M, Frauca E, Undre N; OPTION Study Group. Pharmacokinetics of tacrolimus granules in pediatric de novo liver, kidney, and heart transplantation: The OPTION study. Pediatr Transplant. 2019 Feb;23(1):e13328. doi: 10.1111/petr.13328. Epub 2019 Jan 21. PMID 30665258
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=77